CLINICAL TRIAL: NCT02068131
Title: Phase II Study of Recombinant Anti-tumor and Anti-Virus Protein for Injection Plus Capatabine in Treating Patients With Metastatic Colorectal Cancer After Failure of Standard Treatment
Brief Title: Recombinant Anti-tumor and Anti-virus Protein for Injection Plus Xeloda in Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JH-RC-006
Record Dates: First submitted 2014-02-17; First posted 2014-02-21 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; Novaferon; Recombinant anti-tumor and anti-virus protein for injection; xeloda
MeSH Terms: conditions — Colorectal Neoplasms | interventions — recombinant interferon alpha 2b-like protein; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Novaferon+ xeloda (Experimental): Capecitabine for 2 weeks straight (Days 1-14) followed by 1 week without capecitabine (Days 15-21).
  Recombinant anti-tumor and anti-virus protein for injection(Novaferon), three times per week.
  Interventions: Drug: Novaferon; Drug: Capecitabine

INTERVENTIONS:
Drug: Novaferon — Recombinant anti-tumor and anti-virus protein for injection, 10μg, im, 3 times per week for first 2 weeks, followed by 20μg,im, 3 times per week after 2 weeks.
Drug: Capecitabine — The dose of capecitabine is 1250 mg/m2/dose twice each day, orally, 12 hours apart, for 14 consecutive days, every 21 days (total daily dose = 2500 mg/m2).
  Other Names: Brand name:Xeloda

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-tumor and anti-virus protein for injection plus capecitabine in treating patients with metastatic colorectal cancer who have progressed after standard therapy.

DETAILED DESCRIPTION:
This is a Phase Ⅱ exploratory clinical study. The purpose of this study is to evaluate the efficacy and safety of recombinant anti-tumor and anti-virus protein for injection plus capecitabine in treating patients with metastatic colorectal cancer who have progressed after standard therapy.

All patients will receive recombinant anti-tumor and anti-virus protein for injection and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years.
* Pathologically confirmed metastatic adenocarcinoma of the colon or rectum. All other histological types are excluded.
* Failure of Second-Line and more than second-line treatment, and fluoropyrimidine- and irinotecan- and oxaliplatin-containing regimens.(Subjects who progress during or within 3 months following the last administration of approved standard therapies and terminate standard treatment due to unacceptable toxicity warranting.).If recurrence and metastasis occurred within 6 months after discontinuation of adjuvant chemotherapy, the adjuvant chemotherapy is considered to be first-line treatment.Subject received last-line treatment not including capecitabine.
* At least one measurable lesion according to the RECIST criteria that has not been previously local treated. Minimum indicator lesion size as follows: greater than or equal to 10 mm measured by spiral CT or NMR.Malignant lymph nodes short diameter as follows: greater than or equal to 15 mm measured by spiral CT.
* ECOG performance status 0, 1 or 2.
* Minimum of 4 weeks since any local radiotherapy or surgery for the control of symptoms or severe complications(local radiotherapy for the control of bone metastases is not the limit)，and adequately recovered from toxicities of any prior therapy).
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Prior treatment with novaferon.
* Pregnancy or breast-feeding women or women who may be pregnant were positive drug test before administration.
* Patient of child-bearing potential(male or less than 1 year postmenopausal women) were reluctant to take contraceptive measures.
* Patient who were allergic to Interferon-α or who had interferon-α antibody.
* Patients with uncontrolled central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate(ORR) | every 6 weeks until disease progression,assessed up to 6 months
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.

SECONDARY OUTCOMES:
Disease control rate(DCR) | every 6 weeks until disease progression,assessed up to 6 months
  DCR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments.
Progression-free survival (PFS) | every 6 weeks until disease progression,assessed up to 6 months
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.
Overall survival (OS) | every 8 weeks until death,assessed up to 2 years
  OS is defined as the length of time from random assignment to death or to last contact.
Adverse Events(AEs) | from informed consent form signed to 30 days after termination of administration,assessed up to 6 months
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianming, M.D., Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, China